CLINICAL TRIAL: NCT05302063
Title: A Study to Evaluate the Effect of Spinal Cord Stimulation (SCS) on Clinical Outcomes and Pathology of Painful Diabetic Peripheral Neuropathy (pDPN)
Brief Title: A Study to Evaluate the Effect of Spinal Cord Stimulation (SCS) on Painful Diabetic Peripheral Neuropathy (pDPN)
Acronym: INSPIRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4105
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain
Keywords: Spinal Cord Stimulation; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Spinal Cord Stimulation (SCS) (Experimental): Boston Scientific Spinal Cord Stimulation Systems with multiple modalities
  Interventions: Device: Spinal Cord Stimulation (SCS)

INTERVENTIONS:
Device: Spinal Cord Stimulation (SCS) — Boston Scientific Spinal Cord Stimulation Systems with multiple modalities

SUMMARY:
The purpose of the study is to evaluate the effects of stimulation parameters on clinical outcomes of Spinal Cord Stimulation (SCS) in the treatment of chronic, intractable limb pain resulting from painful Diabetic Peripheral Neuropathy (pDPN).

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of diabetes mellitus, according to International Diabetes guidelines.
* Willing and able to comply with all protocol-required procedures and assessments/evaluations.
* Eligible candidate for SCS from a surgical, cognitive, psychological and psychiatric standpoint per site's routine screening process and based on investigator judgement.
* Subject signed a valid, EC-approved informed consent form (ICF) provided in local language.

Key Exclusion Criteria:

* Primary etiology for lower limb neuropathic pain not due to Diabetic Peripheral Neuropathy (DPN).
* Participating (or intends to participate) in another drug or device clinical trial that may influence the data that will be collected for this study.
* Currently implanted with an active implantable device(s) (e.g., pacemaker, drug pump).
* A female who is pregnant, lactating, or is of childbearing potential and planning to get pregnant during the study or not using adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Pain Relief in Limb Pain | Up to 12 months follow up
  Percent Pain Relief (PPR) in limb pain using a questionnaire where 100% is complete relief and 0% is no relief in pain compared with Baseline

SECONDARY OUTCOMES:
Global Impression of Change | Up to 12 months follow up
  Patient global impression of change (PGI-C) at 3-, 6- and 12-Month Assessment Visit where patients use a seven-point scale to assess how much their condition has improved or worsened relative to their baseline. Subjects will rate themselves as: very much improved; much improved; minimally improved; no change; minimally worse; much worse; or very much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Neuromodulation Corporation
Locations (1):
- Hospital La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No